CLINICAL TRIAL: NCT07316504
Title: Optimal Strategy to Correct Stent underexpAnsion in Resistant Lesions
Acronym: OSCAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2025 SOUTEYRAND
Record Dates: First submitted 2025-09-05; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Coronary Angioplasty; Restenosis; Lithotripsy; Restenosis of Coronary Artery Stent; Angioplasty, Transluminal, Percutaneous Coronary; Percutaneous Coronary Intervention (PCI); OCT Angiography; Optical Coherence Tomography (OCT); Intravascular Lithotripsy; Rotational Atherectomy; OFDI; Intravascular Lithotripsy; Coronary Artery Disease; Coronary Artery Disease (CAD); Coronary Stent Restenosis
Keywords: restenosis; underexpansion; intrastent restenosis; randomized clinical trial; intravascular lithotripsy; baloon PCI; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravascular lithotripsy (Experimental): ISR with UE will be treated by intravascular lithotripsy
  Interventions: Procedure: Intravascular lithotripsy
- Balloon (Active Comparator): ISR with UE will be treated with non compliant balloons, very high-pressure balloons, cutting balloons
  Interventions: Procedure: Balloon

INTERVENTIONS:
Procedure: Intravascular lithotripsy — ISR with UE will be treated by intravascular lithotripsy
  Arms: Intravascular lithotripsy
Procedure: Balloon — ISR with UE will be treated with non compliant balloons, very high-pressure balloons, cutting balloons
  Arms: Balloon

SUMMARY:
Percutaneous coronary intervention (PCI) for in-stent restenosis (ISR) accounts for 5-10% of PCI. ISR may be linked to mechanical complications mainly under-expansion (UE), neointimal hyperplasia and/or neoatherosclerosis. International guidelines recommends non-compliant and very-high-pressure balloons, which lead to sub-optimal angiographic and clinical results. Recently, observational studies have suggested the feasibility and safety of intravascular lithotripsy (IVL) in UE treatment. There are no prospective randomised controlled studies comparing intravascular lithotripsy with balloons in ISR with UE.

DETAILED DESCRIPTION:
In-stent restenosis (ISR) angioplasties account for between 5 and 10% of Percutaneous coronary intervention (PCI). Several mechanisms are causing RIS, including neointimal hyperplasia, neoatherosclerosis, and/or mechanical complications, mainly stent under-expansion. In addition, the calcified lesions associated with stent under-expansion are under-diagnosed in angiography as shown by intra-coronary imaging studies. The stent under-expansion is defined as a ratio between the minimum intrastent surface area and the average vessel lumen of <80%. Currently, the management of these lesions is not codified and consists empirically of the use of non-compliant balloons, cutting balloons, and/or very high-pressure balloons. These treatments result in suboptimal angiographic results, with clinical consequences in terms of revascularization recurrence (angina, unstable angina, and in 25% of cases, acute coronary syndrome).

A growing interest in intravascular lithotripsy (IVL) use to treat these calcified lesions with stent underexpansion appears as an appealing option for a safe procedure but without robust data on efficacy. Furthermore, guidelines published in 2020 by the expert consensus of the EAPCI (European Association of Percutaneous Coronary Interventions) classified IVL among the therapeutic strategy indicated in stent under-expansion with calcified lesions. The OSCAR study is a randomized, controlled, multicenter trial investigating the use of IVL compared to other standard strategies in the treatment of in-stent restenosis with under-expansion.

ELIGIBILITY:
Inclusion criteria :

* Patient who have undergone coronary angiography with ISR, defined as ≥50% reduction of the diameter of the intrastent lumen occurring ≥ 6 months after stent implantation
* And with a suspicion of stent under-expansion on angiography, possibly assisted by a stent enhancement technique
* The reference diameter of the target vessel must be ≥2.5 mm and ≤5.0 mm.
* Coronary flow must be TIMI 3
* Ability to cross the lesion with the OCT catheter (possibly after predilatation with a balloon up to 2 mm)
* Patient affiliated to the French National Health Insurance

Exclusion criteria :

* Heart failure with NYHA III or IV (or cardiogenic shock)
* LVEF <20%
* Chronic renal failure with clearance <30mL/mn according to CKD
* Pregnant or breast-feeding women
* Patient with a condition/comorbidity that could reduce compliance with the protocol, including pre-specified study follow-up
* Patient participating in another ongoing medical study evaluating a pharmacological or biological agent or medical device, unless authorized by the concomitant protocol.
* Patient unable to tolerate double antiaggregation (i.e., aspirin and clopidogrel or prasugrel or ticagrelor) for at least 6 months.
* Possible or defined thrombus (by angiography or endovascular imaging) in the target vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Post PCI Stent expansion | At enrollment
  Minimal stent area (MSA)/average reference vessel area

SECONDARY OUTCOMES:
Minimal stent area >4.5mm2 or Stent expansion ≥80% | At enrollment
  Number of patients with Efficiency (yes/no) Efficiency defined by: optimal stent expansion (Minimal Stent Area [MSA]/mean reference vessel diameter ≥ 80%) and/or MSA > 4.5 mm².
Successful lithotripsy catheter delivery | At enrollment
  Number of patients with successful lithotripsy catheter delivery
Procedural success evaluated by the occurence of the clinical events below | Day 1 - Day 7
  Procedural success is defined as residual stenosis < 50% or MSA > 4.5 mm2 and no angiographic complications (i.e., acute dissection (types B to F), perforation, acute vessel obstruction, persistent slow flow, or no reflow) or distal embolization.
  * Residual stenosis < 50% post-procedure (assessed by Quantitative Coronary Angiography (QCA))
  * No significant stent malapposition
  * Target lesion failure defined as: cardiac death, myocardial infarction (unless clearly attributable to a vessel other than the target vessel) and target lesion revascularization (TLR) during index hospitalization (Day 1-Day 7).
  * Target Vessel Failure (TVF) defined as: cardiac death, myocardial infarction (unless clearly attributable to a vessel other than the target vessel) and target vessel revascularization (TVR) during index hospitalization (Day 1-Day 7).
Peri-procedural complications evaluated by the occurence of the clinical events below | Day 1- Day 7
  * Coronary arteries: Dissection (A-F), persistent slow flow, no reflow, perforation, embolization, acute vessel occlusion, side branch occlusion (>1.5 mm, final TIMI flow)
  * Peri-procedural infarction
  * Vascular access complications: dissection, hematoma, pseudoaneurysm, hemorrhage
  * Radiation protection parameters: procedure time (min), air kerma, total dose-area product (DAP), iodine quantity (ml)
Safety criteria evaluated by the occurence of the clinical events below | From enrollment to the end of study at Month 36
  * All-cause mortality
  * Cardiovascular mortality
  * Peri-procedural myocardial infarction
  * Spontaneous myocardial infarction
  * Probable or definite stent thrombosis
  * Stroke
  * Major bleeding
Efficiency criteria evaluated by any of the clinical events described below | From enrollment to the end of study at Month 36
  * Target Lesion Revascularization (TLR)
  * Target Vessel Revascularization (TVR)
  * Target Vessel Non-Target lesion Revascularization (TV-NTLR)
  * Non-Target Vessel Revascularization (NTVR)
  * Any hospitalization (for cardiac reasons or related to the procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Géraud Souteyrand, MD, PhD, Principal Investigator — CHU de Clermont-Ferrand
Locations (2):
- France (2):
  - Clermont Ferrand Hospital, Clermont-Ferrand, Auvergne
  - CHU de Clermont-Ferrand, Clermont-Ferrand

IPD SHARING:
Plan to Share IPD: No